CLINICAL TRIAL: NCT03379792
Title: The Influence of Glycemic Control and Obesity on Energy Balance and Metabolic Flexibility in Type 1 Diabetes
Acronym: ACME
Status: Completed | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMDFH 1144866
Record Dates: First submitted 2017-11-15; First posted 2017-12-20 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes
Keywords: Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Type 1 Diabetes: BMI Classified as Lean: Participants with type 1 diabetes with a BMI between 18.0-24.9 kg/m^2.
- Type 1 Diabetes: BMI Classified as Overweight: Participants with type 1 diabetes with a BMI between 25.0-29.9 kg/m^2.
- Type 1 Diabetes: BMI Classified as Obese: Participants with type 1 diabetes with a BMI between 30.0-39.9 kg/m^2.
- Control: BMI Classified as Lean: Control participants without diabetes with a BMI between 18.0-24.9 kg/m^2.
- Control: BMI Classified as Overweight: Control participants without diabetes with a BMI between 25.0-29.9 kg/m^2.
- Control: BMI Classified as Obese: Control participants without diabetes with a BMI between 30.0-39.9 kg/m^2.

SUMMARY:
The purpose of this study is to measure the metabolic phenotype of a range of body weights in individuals with and without type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 19 to 30 years of age, inclusive.
2. Type 1 Diabetes Cohort:

   1. Diagnosis of type 1 diabetes for greater than 1 year at screening.
   2. Hemoglobin A1c 6.5-13% or

   Control Cohort Without Diabetes:

   a. Healthy individuals without diabetes matched to T1D cohort by BMI and gender
3. Able to provide informed consent.
4. BMI 18-39.9 kg/m^2

Exclusion Criteria:

1. Type 2 diabetes
2. History or presence of cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, clinically significant abnormalities on EKG, presence of cardiac pacemaker, implanted cardiac defibrillator)
3. Liver disease (AST or ALT >2.5 times the upper limit of normal), history of hepatitis
4. Kidney disease (creatinine >1.6 mg/dl or estimated glomerular filtration rate (GFR)<60 ml/min)
5. Dyslipidemia, including triglycerides >800 mg/dl, LDL >200 mg/dl
6. Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women)
7. Thyroid dysfunction (suppressed thyroid-stimulating hormone (TSH), elevated TSH <10 µIU/ml if symptomatic or elevated TSH >10 µIU/ml if asymptomatic)
8. Uncontrolled hypertension (BP >160 mmHg systolic or > 100mmHg diastolic)
9. History of cancer within the last 5 years (skin cancers, with the exception of melanoma, may be acceptable).
10. Initiation or change in hormone replacement therapy within the past 3 months (including, but not limited to thyroid hormone, birth control or estrogen replacement therapy)
11. History of organ transplant
12. History of HIV, active Hepatitis B or C, or Tuberculosis
13. Pregnancy, lactation or 6 months postpartum from screening visit
14. History of major depression
15. Psychiatric disease prohibiting adherence to study protocol
16. History of eating disorders
17. Cushing's disease or syndrome
18. History of bariatric surgery
19. Tobacco use within the past 3 months
20. History of drug or alcohol abuse (≥3 drinks per day) within the last 5 years
21. Use of oral or injectable anti-hyperglycemic agents (except insulin)
22. Current use of beta-adrenergic blocking agents
23. Use of antibiotics within the past 3 months
24. Weight >450 lbs (This is DEXA table weight limit)
25. Metal implants (pace-maker, aneurysm clips) based on Investigator's judgment at screening
26. Unable to participate in MRI or magnetic resonance spectroscopy (MRS) assessment based on Investigator's judgment at screening
27. Participants with strict dietary concerns (e.g. vegetarian or kosher diet, multiple food allergies, or allergies to food we will provide them during the study)
28. Gastrointestinal disorders including: inflammatory bowel disease or malabsorption, swallowing disorders, suspected or known strictures, fistulas or physiological/mechanical GI obstruction, history of gastrointestinal surgery, Crohn's disease or diverticulitis.
29. Presence of any condition that, in the opinion of the investigator, compromises participant safety or data integrity or the participant's ability to complete study visits

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults with type 1 diabetes diagnosed greater than or equal to 1 year prior to screening, or control young adults without diabetes, both within a range of BMI classifications (18-39.9 kg/m^2).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes; Elizabeth Mayer-Davis, PhD, Principal Investigator — UNC Chapel Hill; David M Maahs, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Chillaron JJ, Benaiges D, Mane L, Pedro-Botet J, Flores Le-Roux JA. Obesity and type 1 diabetes mellitus management. Minerva Endocrinol. 2015 Mar;40(1):53-60. Epub 2014 Nov 21. PMID 25413942
- [Background] Maahs DM, Ogden LG, Dabelea D, Snell-Bergeon JK, Daniels SR, Hamman RF, Rewers M. Association of glycaemia with lipids in adults with type 1 diabetes: modification by dyslipidaemia medication. Diabetologia. 2010 Dec;53(12):2518-25. doi: 10.1007/s00125-010-1886-6. Epub 2010 Sep 4. PMID 20820753
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group; Nathan DM, Zinman B, Cleary PA, Backlund JY, Genuth S, Miller R, Orchard TJ. Modern-day clinical course of type 1 diabetes mellitus after 30 years' duration: the diabetes control and complications trial/epidemiology of diabetes interventions and complications and Pittsburgh epidemiology of diabetes complications experience (1983-2005). Arch Intern Med. 2009 Jul 27;169(14):1307-16. doi: 10.1001/archinternmed.2009.193. PMID 19636033
- [Background] Jacob AN, Salinas K, Adams-Huet B, Raskin P. Potential causes of weight gain in type 1 diabetes mellitus. Diabetes Obes Metab. 2006 Jul;8(4):404-11. doi: 10.1111/j.1463-1326.2005.00515.x. PMID 16776747
- [Background] Rigalleau V, Lasseur C, Pecheur S, Chauveau P, Combe C, Perlemoine C, Baillet L, Gin H. Resting energy expenditure in uremic, diabetic, and uremic diabetic subjects. J Diabetes Complications. 2004 Jul-Aug;18(4):237-41. doi: 10.1016/S1056-8727(03)00077-1. PMID 15207844
- [Background] Carlson MG, Campbell PJ. Intensive insulin therapy and weight gain in IDDM. Diabetes. 1993 Dec;42(12):1700-7. doi: 10.2337/diab.42.12.1700. PMID 8243815
- [Background] Greco AV, Tataranni PA, Mingrone G, De Gaetano A, Manto A, Cotroneo P, Ghirlanda G. Daily energy metabolism in patients with type 1 diabetes mellitus. J Am Coll Nutr. 1995 Jun;14(3):286-91. doi: 10.1080/07315724.1995.10718509. PMID 8586779
- [Background] Nair KS, Halliday D, Garrow JS. Increased energy expenditure in poorly controlled Type 1 (insulin-dependent) diabetic patients. Diabetologia. 1984 Jul;27(1):13-6. doi: 10.1007/BF00253494. PMID 6147290
- [Derived] Casu A, Nunez Lopez YO, Yu G, Clifford C, Bilal A, Petrilli AM, Cornnell H, Carnero EA, Bhatheja A, Corbin KD, Iliuk A, Maahs DM, Pratley RE. The proteome and phosphoproteome of circulating extracellular vesicle-enriched preparations are associated with characteristic clinical features in type 1 diabetes. Front Endocrinol (Lausanne). 2023 Jul 28;14:1219293. doi: 10.3389/fendo.2023.1219293. eCollection 2023. PMID 37576973
- [Derived] Corbin KD, Igudesman D, Addala A, Casu A, Crandell J, Kosorok MR, Maahs DM, Pokaprakarn T, Pratley RE, Souris KJ, Thomas JM, Zaharieva DP, Mayer-Davis EJ; ACT1ON Consortium. Design of the Advancing Care for Type 1 Diabetes and Obesity Network energy metabolism and sequential multiple assignment randomized trial nutrition pilot studies: An integrated approach to develop weight management solutions for individuals with type 1 diabetes. Contemp Clin Trials. 2022 Jun;117:106765. doi: 10.1016/j.cct.2022.106765. Epub 2022 Apr 20. PMID 35460915
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 1 Diabetes: BMI Classified as Lean: Participants with type 1 diabetes who had a BMI between 18.0-24.9 kg/m^2.
Period: Overall Study
Arm/Group | Type 1 Diabetes: BMI Classified as Lean | Type 1 Diabetes: BMI Classified as Overweight | Type 1 Diabetes: BMI Classified as Obese | Control: BMI Classified as Lean | Control: BMI Classified as Overweight | Control: BMI Classified as Obese
Started | 6 | 9 | 5 | 4 | 4 | 4
Completed | 6 | 9 | 5 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 1 Diabetes: BMI Classified as Lean | Type 1 Diabetes: BMI Classified as Overweight | Type 1 Diabetes: BMI Classified as Obese | Control: BMI Classified as Lean | Control: BMI Classified as Overweight | Control: BMI Classified as Obese | Total
Number analyzed (Participants) | 6 | 9 | 5 | 4 | 4 | 4 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (1.9) | 24.6 (3.2) | 25.8 (3.5) | 24.3 (3.3) | 24.0 (2.1) | 27.8 (6.1) | 24.6 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 3 | 1 | 1 | 15
  Male | 2 | 5 | 3 | 1 | 3 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 1 | 1 | 2 | 2 | 14
  Not Hispanic or Latino | 3 | 3 | 4 | 2 | 2 | 2 | 16
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 2 | 1 | 1 | 1 | 6
  White | 5 | 6 | 3 | 2 | 3 | 3 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 5 | 4 | 4 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Energy Expenditure
Description: Measured via whole room calorimetry; based on oxygen consumption and carbon dioxide production measured using gas analyzers, as well as 14-hour urinary nitrogen excretion; calculated using established equations.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Kilocalories
Arm/Group | Type 1 Diabetes: BMI Classified as Lean | Type 1 Diabetes: BMI Classified as Overweight | Type 1 Diabetes: BMI Classified as Obese | Control: BMI Classified as Lean | Control: BMI Classified as Overweight | Control: BMI Classified as Obese
Number analyzed (Participants) | 6 | 9 | 5 | 3 | 3 | 3
Kilocalories | 1978.3 (337.8) | 1969.8 (236.3) | 2414.8 (419.1) | 1497.7 (123.6) | 1902.0 (406.0) | 2671.3 (402.7)
Statistical Analysis 1: Comparison: Type 1 Diabetes: BMI Classified as Lean vs Control: BMI Classified as Lean; Test type: Other; p = 0.24, t-test, 2 sided
Statistical Analysis 2: Comparison: Type 1 Diabetes: BMI Classified as Overweight vs Control: BMI Classified as Overweight; Test type: Other; p = 0.22, t-test, 2 sided
Statistical Analysis 3: Comparison: Type 1 Diabetes: BMI Classified as Obese vs Control: BMI Classified as Obese; Test type: Other; p = 1.0, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 28-42 days
Arm/Group | Type 1 Diabetes: BMI Classified as Lean | Type 1 Diabetes: BMI Classified as Overweight | Type 1 Diabetes: BMI Classified as Obese | Control: BMI Classified as Lean | Control: BMI Classified as Overweight | Control: BMI Classified as Obese
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/5 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/5 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/6 | 5/9 | 1/5 | 0/4 | 0/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 1 Diabetes: BMI Classified as Lean (N=6) | Type 1 Diabetes: BMI Classified as Overweight (N=9) | Type 1 Diabetes: BMI Classified as Obese (N=5) | Control: BMI Classified as Lean (N=4) | Control: BMI Classified as Overweight (N=4) | Control: BMI Classified as Obese (N=4)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT03379792/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT03379792/ICF_002.pdf